CLINICAL TRIAL: NCT00402805
Title: Improving the Humoral Response to Influenza Vaccine in Lung Transplant Recipients by an Intradermal Strategy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06-0380-AE
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2006-11

CONDITIONS: Lung Transplantation; Influenza Vaccines
Keywords: Influenza vaccine; Intradermal; Lung transplantation
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Trivalent Inactivated Influenza Vaccine

SUMMARY:
The purpose of this study is to test the specific humoral response after an intramuscular and intradermal influenza vaccination in lung transplant recipients

DETAILED DESCRIPTION:
Influenza virus is an important cause of morbidity in the lung transplant population and can lead to viral and bacterial pneumonia and contribute to the bronchiolitis obliterans syndrome. Although the annual influenza vaccine is recommended for lung transplant patients, studies have shown that a single intramuscular (i.m.) dose has poor immunogenicity. There are no studies that define the effect of intradermal doses in this population. We plan to study the immunogenicity of a two-dose regimen of influenza vaccine in 50 lung transplant patients during the 2006-2007 season. After the initial i.m. injection, a second dose will be given intradermally 4 weeks later. Antibody titers will be evaluated by a standard hemagglutination inhibition assay. We hypothesize that the second dose intradermally will significantly increase the proportion of vaccine responders.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipients greater than 3 months post-transplant

Exclusion Criteria:

* · Egg allergy

  * Previous life-threatening reaction to influenza vaccine (ie Guillain Barre Syndrome)
  * On anticoagulants such as warfarin that precludes intramuscular injection
  * Ongoing therapy for rejection
  * Febrile illness in the past two weeks
  * Unable to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
HIA titers 4 weeks after influenza vaccination

SECONDARY OUTCOMES:
Local and systemic adverse events to vaccination and rates
of allograft rejection in the 6 months following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Multi-Organ Transplant Program, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Soesman NM, Rimmelzwaan GF, Nieuwkoop NJ, Beyer WE, Tilanus HW, Kemmeren MH, Metselaar HJ, de Man RA, Osterhaus AD. Efficacy of influenza vaccination in adult liver transplant recipients. J Med Virol. 2000 May;61(1):85-93. PMID 10745238
- [Background] Mazzone PJ, Mossad SB, Mawhorter SD, Mehta AC, Schilz RJ, Maurer JR. The humoral immune response to influenza vaccination in lung transplant patients. Eur Respir J. 2001 Dec;18(6):971-6. doi: 10.1183/09031936.01.00215201. PMID 11829104
- [Background] Belshe RB, Newman FK, Cannon J, Duane C, Treanor J, Van Hoecke C, Howe BJ, Dubin G. Serum antibody responses after intradermal vaccination against influenza. N Engl J Med. 2004 Nov 25;351(22):2286-94. doi: 10.1056/NEJMoa043555. Epub 2004 Nov 3. PMID 15525713
- [Background] Vilchez RA, McCurry K, Dauber J, Lacono A, Griffith B, Fung J, Kusne S. Influenza virus infection in adult solid organ transplant recipients. Am J Transplant. 2002 Mar;2(3):287-91. doi: 10.1034/j.1600-6143.2002.20315.x. PMID 12096793